CLINICAL TRIAL: NCT03550950
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of JNJ-64232025 in Healthy Participants
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of JNJ-64232025 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CR108448; 2017-003986-82 (EudraCT Number); 64232025ARA1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-05-29; First posted 2018-06-11 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Ascending Dose (SAD) IV Cohort (Experimental): Participants will receive single intravenous (IV) dose of JNJ-64232025 or placebo in Cohorts 1 to 6 on Day 1.
  Interventions: Drug: JNJ-64232025 IV; Drug: Placebo
- Subcutaneous (SC) Cohort (Experimental): Participants will receive single dose of JNJ-64232025 or placebo as SC injection.
  Interventions: Drug: JNJ-64232025 SC; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-64232025 IV — JNJ-64232025 will be administered as IV infusion.
  Arms: Single Ascending Dose (SAD) IV Cohort
Drug: JNJ-64232025 SC — JNJ-64232025 will be administered as SC injection.
  Arms: Subcutaneous (SC) Cohort
Drug: Placebo — Matching placebo will be administered as IV infusion or SC injection.

SUMMARY:
The purpose of this study is to assess the safety and tolerability of JNJ-64232025 following single ascending intravenous (IV) study intervention administrations and a single subcutaneous (SC) intervention administration in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of non-childbearing potential (postmenopausal or permanently sterile)
* Have a body mass index (BMI) between 19 and 30 kilogram per meter square (kg/m^2) (BMI = weight/height^2), and a body weight of 50 to 100 kilogram (kg), inclusive
* Healthy on the basis of medical history, a physical examination, vital signs, and 12 lead electrocardiogram (ECG) performed at screening
* Healthy on the basis of clinical laboratory tests performed at screening and Day -1
* A woman must have a negative highly sensitive serum pregnancy test at screening and a negative urine pregnancy test on Day -1

Exclusion Criteria:

* Has history of any clinically significant medical illness or medical disorders the investigator considers should exclude the participant, including (but not limited to), neuromuscular, hematological disease, immune deficiency state, respiratory disease, hepatic or gastrointestinal disease, neurological or psychiatric disease, ophthalmological disorders, neoplastic disease, renal or urinary tract diseases, or dermatological disease
* Has a disease or disease treatment associated with immune suppression or lymphopenia, these include but are not limited to bone marrow or organ transplantation, lymphoproliferative disorders, T- or B-cell deficiency syndromes, splenectomy, functional asplenism, and chronic granulomatous disease
* Has a personal history of or conditions associated with thromboembolic events or bleeding disorders, including (but not limited to) myocardial infarction (MI), cerebral vascular accident (CVA)/stroke, deep vein thrombosis (DVT), pulmonary embolism (PE), hemophilia, or menometrorrhagia
* Has history of allergy or adverse reactions to shellfish, aluminum, aluminum hydroxide keyhole limpet hemocyanin (KLH), tetanus or tetanus toxoid or its excipients
* Has a known or suspected intolerance or hypersensitivity to any biologic medication or known allergies or clinically significant reactions to murine, chimeric, or human proteins, monoclonal antibodies or antibody fragments, or to any components of the formulation of JNJ-64232025 and its excipients used in this study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2019-02-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAE) by Severity | Up to Day 113
  An adverse event (AE) is any untoward medical occurrence in a participant who receive study drug without regard to possibility of causal relationship. The severity of the TEAEs will be assessed as mild, moderate, or severe.
Number of Participants with Serious Adverse Events (SAE) | Up to Day 113
  An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Number of Participants with Clinically Significant Changes in Vital Signs | Up to Day 113
  Number of participants with clinically significant changes in the vital signs including temperature, pulse/heart rate, respiratory rate, and blood pressure will be reported.
Number of Participants with ECG Abnormalities | Up to Day 113
  Number of participants with electrocardiogram (ECG) abnormalities will be reported.
Number of Participants with Clinical Laboratory Abnormalities | Up to Day 113
  Number of participants with clinical laboratory abnormalities, including cytomegalovirus (CMV) and Epstein-Barr virus (EBV) viral loads, will be reported.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of JNJ-64232025 | Up to Day 113
  The Cmax is the maximum observed plasma concentration of JNJ-64232025.
Time to Reach Maximum Observed Plasma Concentration (Tmax) of JNJ-64232025 | Up to Day 113
  The Tmax is defined as actual sampling time to reach maximum observed plasma concentration of JNJ-64232025.
Area Under the Plasma Concentration-Time Curve from Time Zero to Infinity with Extrapolation of the Terminal Phase (AUC[0-infinity]) | Up to Day 113
  The AUC(0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(0-last) and C(0-last)/lambda(z); wherein AUC(0-last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(0-last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Area Under the Plasma Concentration-Time Curve from Time Zero to the Time Corresponding to the Last Quantifiable Concentration (AUC[0-last]) | Up to Day 113
  The AUC(0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time.
Terminal Half-Life (t1/2) | Up to Day 113
  The t1/2 is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Total Systemic Clearance (C/L) | Up to Day 113
  Systemic clearance is a quantitative measure of the rate at which a drug substance is removed from the body. The total systemic clearance after intravenous dose was estimated by dividing the total administered dose by the plasma AUC(0-infinity).
Apparent Total Systemic Clearance After Extravascular Administration (CL/F) | Up to Day 113
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. CL/F is the apparent total systemic clearance after extravascular administration.
Volume of Distribution Based on Terminal Phase (Vz) | Up to Day 113
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug.
Apparent Volume of Distribution Based on Terminal Phase After Extravascular Administration (Vz/F) | Up to Day 113
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug. Apparent volume of distribution after subcutaneous dose (Vz/F) is influenced by the fraction absorbed.
Relative SC Bioavailability (F%) | Up to Day 113
  Relative SC bioavailability will be calculated using the following equation: F (%[percent]) = AUC(0-infinity),SC/ mean AUC(0-infinity),IV *100%.
Number of Participants with Anti-JNJ 64232025 Antibodies | Up to Day 113
  Number of participants with anti-JNJ-64232025 antibodies will be assessed.
Number of Participants with Anti-KLH and Anti-Tetanus Antibodies | Up to Day 113
  Number of participants with antibodies to anti-Keyhole Limpet Hemocyanin (KLH) and anti-tetanus will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- SGS Life Science Services, Antwerp, Belgium